CLINICAL TRIAL: NCT03254264
Title: Impact of Early Intervention on Neurocognitive Profile of Children With Autism Spectrum Disorder
Brief Title: Impact of Early Interventions on Neurocognitive Profile of Children With Autism Spectrum Disorder
Acronym: IDEAEYE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: one inclusion and not others
Sponsor: Hôpital le Vinatier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-A00696-43
Record Dates: First submitted 2017-08-16; First posted 2017-08-18 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: ESDM is a comprehensive relational, developmental and behavioral intervention. It's described in a manual for professional (Rogers et al, 2010).
  Children receive ESDM at minimum 12H per week by trained therapist. Therapist work in collaboration with parents (at home) and preschool or nursery.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESDM-12 (Experimental): an experimental group of 60 children receiving 12 hours a week of Early Start Denver Model (ESDM) intervention delivered by trained therapists during 2 years ESDM is a comprehensive relational, developmental and behavioral intervention.It's described in a manual for Professional and parents.
  Interventions: Behavioral: Early Start Denver Model
- Control group (Active Comparator): a control group of 120 children receiving typical heterogeneous 'as-usual' intervention proposed by professionals and public services over the same period.
  Interventions: Behavioral: 'as-usual' intervention

INTERVENTIONS:
Behavioral: Early Start Denver Model — ESDM is a comprehensive relational, developmental and behavioral intervention. It's described in a manual for professional (Rogers et al, 2010).
  Children receive ESDM at minimum 12H per week by trained therapist. Therapist work in collaboration with parents (at home) and preschool or nursery.
  Arms: ESDM-12
Behavioral: 'as-usual' intervention — a control group receiving typical heterogeneous 'as-usual' intervention proposed by professionals and public services over the same period.
  Arms: Control group

SUMMARY:
The Early start Denver model (Rogers, 2010; Dawson, 2010) is a developmental and behavioral model that aim to enhance socio-comunicative abilities and also global development of children with Autism spectrum disorder (ASD). The purpose of this study is to identify changes in neurocognitive profile of children population with ASD receiving Early Start Denver Model (ESDM) applied 12 hours per week in comparison to children receiving other interventions. That is a study proposed to children with ASD and their families that participate already to a randomized control study called IDEA registered on clinicaltrials.gov NCT02608333.

the investigators hypothesized that ESDM would increase social cognition, reduce shifting attention time and increase preference for unpredictable stimuli.

DETAILED DESCRIPTION:
IDEA is a multicenter (4 centers in France and 1 center in Belgium), randomized, controlled, single blind trial using a modified Zelen design .It concerns children with ASD aged 15 to 36 months without severe neurological or physical disorder and living in the proximity of one the early intervention units. After diagnostic, Children will be included in a longitudinal cohort with the consent of the parents. Sixty children will be drawn lots among 180 children of the cohort and will be included in an ESDM intervention with the consent of the parents. Two groups will be compared: an experimental group of 60 children receiving 12 hours a week of ESDM intervention delivered by trained therapists during 2 years and a control group of 120 children receiving typical heterogeneous 'as-usual' intervention proposed by professionals and public services over the same period. In IDEA development of communication and social interactions and global developmental of all the children will be measured at different time points (at baseline (t0), after 1 year (t1), after 2 years( t2)) over the two years through standardized tests such as Autism diagnostic observation Schedule (ADOS-2), Mullen Scales of Early Learning (MSEL) and the Vineland Adaptive Behavior Scale (VABS-2).

Children will be included in this second study called IDEA-EYE with parents' consent. Then, preference for biological motion and social scene, shifting attention time and preference for sameness will be measure in both groups with an Eye-tracker Tobii TX 300 at t0,t1 and t2. These measures will also be collected in a group of children without ASD at t0,t1 and t2.

the investigators expect, as primary criteria, a significant superior time spend on biological motion in ESDM group versus control group after 2 years of treatment. the investigators also expect a significant superior orientation toward eyes in complex social scenes, an inferior shifting attention time and a superior preference for unpredictable stimuli in ESDM group versus ASD control group after 2 years. the investigators also expect that ESDM group would have time spend on biological motion, orientation toward eyes in complex scenes, shifting attention time and preference for unpredictable stimuli comparable to children without ASD after 2 years.

This study would allow better understanding of ESDM active principles.

ELIGIBILITY:
Inclusion Criteria:

* Children 15 months to 36 months
* Children with autism spectrum disorder (according to international criteria, ADI and ADOS)
* DQ at 30 at least at the Early Learning Mullen Scale
* Family domiciled within 40 minutes of an early intervention unit

Exclusion Criteria:

* Severe neurological or physical disorder identified in the child or family that would interfere with intervention
* Unavailability of the family for regular monitoring of the child by the investigator center
* Child with a Rett Sd or Childhood disintegrative disorders
* Visual problems or with eyes in general

Ages: 15 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2017-05-29 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the time spent on biological motion in the task of visual preference stimuli. | 2 years
  2 different types of stimuli (dynamic biological or geometrical movements) are presented in parallel on each part of the screen alternatively (left and/ or right). Child sit at 60 cm from the screen of the Eye-tracker can look towards the one or the other one stimuli.

SECONDARY OUTCOMES:
Average proximity from pattern eyes norm in complex social scene task | 2 years
  A 3-minute cartoon is displayed on a Tobii TX 300 eye-tracker. Inspired by the concept of a heatmap, for each frame of the video "normative" gaze pattern distribution are created by employing kernel density distribution estimation on the raw gaze data of TD individuals (Botev et al., 2009). For each patient we then will calculate the "distance" of his/hers gaze coordinates from this "norm". Thus we will obtain one measure per frame of Proximity from the "norm", which will be then averaged for the duration of the video.
Difference of saccadic latencies between overlap and gap condition | 2 years
  in a gap/ overlap paradigm displayed on the Tobii TX 300 eye-tracker screen, we will measure the difference of mean of saccadic latencies between the two conditions.
Time spent on unpredictable stimuli | 2 years
  2 type of stimuli are presented on the Eye-tracker screen : one very predictable stimuli and unpredictable stimuli.

CONTACTS AND LOCATIONS:
Overall Officials: GEOFFRAY Marie-Maude, PHD, Principal Investigator — Centre Hospitalier le Vinatier
Locations (1):
- Hopital Vinatier, Bron, France